CLINICAL TRIAL: NCT04493554
Title: The Effects of Vasopressin on Attention Control: An Eye-tracking Study
Brief Title: The Effects of Vasopressin on Attention Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-70
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Healthy
MeSH Terms: interventions — Vasopressins

STUDY DESIGN:
Intervention Model Description: Between-subject randomized placebo-controlled double-blind pharmacological eye-tracking design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vasopressin (Experimental): Vasopressin (20 IU) intranasally
  Interventions: Drug: Vasopressin
- Placebo (Placebo Comparator): Placebo intranasally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vasopressin — Administration of vasopressin (20 IU) intranasally
  Arms: Vasopressin
Drug: Placebo — Administration of placebo intranasally
  Arms: Placebo

SUMMARY:
The main aim of the present study is to investigate whether intranasal vasopressin (20IU) could influence attention control in a social-emotional saccade/antisaccade eye-tracking paradigm.

DETAILED DESCRIPTION:
A number of previous studies have reported vasopressin's effect on human social behavior and social cognition, although it remains unclear whether vasopressin could modulate attention allocation including stimulus-driven bottom-up control and goal-directed top-down control. In the current randomized, between-subject, placebo controlled study, 89 healthy male subjects will be recruited and receive either vasopressin (20 IU) or placebo control administered intranasally. 45 minutes after treatment subjects will be required to complete a social-emotional saccade /antisaccade eye-tracking paradigm. The paradigm uses social (happy, sad, angry, fear, and neutral faces) as well as non-social (oval shapes) stimuli to explore social- and emotion-specific effects of vasopressin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants
* Non smokers

Exclusion Criteria:

* Previous or current medical, psychiatric, neurological disorder
* Regular medication
* Use of any psychoactive substances in the 24 hours before experiment
* Contra-indications for vasopressin
* Contra-indications for eye-tracking data acquisition

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Effect of vasopressin administration on saccade/antisaccade latencies towards social (facial) versus non-social (shape) stimuli | 45 minutes - 100 minutes after treatment
  Comparison between social-specific saccade/antisaccade latencies (in milliseconds) between the vasopressin and placebo treatment conditions
Effect of vasopressin administration on error rates of saccade/antisaccade for social (facial) versus non-social (shape) stimuli | 45 minutes - 100 minutes after treatment
  Comparison between social-specific error rates of saccade/antisaccade between the vasopressin and placebo treatment conditions

SECONDARY OUTCOMES:
Emotion-specific effects of vasopressin administration on saccade/antisaccade latencies towards the separate facial emotions | 45 minutes - 100 minutes after treatment
  Comparison between emotion-specific saccade/antisaccade latencies (in milliseconds) between the vasopressin and placebo treatment conditions
Emotion-specific effects of vasopressin administration on saccade/antisaccade error rates for the separate facial emotions | 45 minutes - 100 minutes after treatment
  Comparison between emotion-specific saccade/antisaccade error rates between the vasopressin and placebo treatment conditions

CONTACTS AND LOCATIONS:
Overall Officials: Keith Kendrick, PhD, Principal Investigator — University of Electronic Science and Technology of China (UESTC)
Locations (1):
- University of Electronic Science and Technology of China(UESTC), Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No